CLINICAL TRIAL: NCT07049653
Title: A Non-Interventional Multi-Database Post-Authorisation Study to Assess Pregnancy-Related Safety Data From Women With SLE Exposed to Anifrolumab
Brief Title: Anifrolumab Pregnancy Study
Acronym: ROSE
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461R00028
Record Dates: First submitted 2025-05-23; First posted 2025-07-03 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: pregnancy, anifrolumab, SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Exposed cohort: Pregnant individuals with a diagnosis of SLE who are exposed to anifrolumab at any time during pregnancy
- Unexposed cohort: Pregnant individuals with a diagnosis of moderate/severe SLE who are not exposed to anifrolumab at any time during pregnancy but who are exposed to other products for the treatment of SLE

SUMMARY:
This is a non-interventional multi-database post-authorisation study to assess pregnancy-related safety data from women with SLE exposed to Anifrolumab.

DETAILED DESCRIPTION:
The aim of this study is to describe congenital malformations, adverse pregnancy and birth outcomes in pregnancies/offspring from women with moderate/severe SLE exposed to anifrolumab during pregnancy and to compare with outcomes in women with moderate/severe SLE who are exposed to other standard of care but not anifrolumab. Adverse outcomes related to infant growth up to one year of age will also be investigated.

ELIGIBILITY:
Inclusion criteria for EXPOSED SOURCE POPULATION:

* Women with a continuous enrolment in the database for ≥ 12 months prior to LMP2
* Women diagnosed with SLE before pregnancy
* Women exposed to anifrolumab (polytherapy, added to SLE SOC) during pregnancy and/or 16-week period prior to LMP2

Exclusion criteria for EXPOSED SOURCE POPULATION:

- Pregnancies whose date of conception cannot be established

Inclusion criteria for UNEXPOSED SOURCE POPULATION:

* Women with a continuous enrolment in the database for ≥ 12 months prior to LMP2
* Women diagnosed with SLE before pregnancy
* Women treated with SLE SOC during pregnancy

Exclusion criteria for UNEXPOSED SOURCE POPULATION:

* Women treated with anifrolumab during pregnancy and/or 16-week period prior to LMP2
* Pregnancies whose date of conception cannot be established

Inclusion criteria for EXPOSED and UNEXPOSED STUDY POPULATION:

- Women with moderate/severe SLE

Exclusion criteria for EXPOSED and UNEXPOSED STUDY POPULATION:

* Women with a history of CM or chromosomal abnormalities (according to available records), before delivery
* Women prescribed a confirmed teratogenic drug prior to LMP2 with a time period of 5-half-lives of relevant drug or during pregnancy

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will encompass women with SLE of child-bearing potential age (15-49 years old) who start anifrolumab or other selected SLE treatments.
  For the safety outcomes analyses the study population will include pregnant women and their infant born anytime during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 627 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2030-12-10 (Estimated); Study Completion 2030-12-10 (Estimated)

PRIMARY OUTCOMES:
Risk of major congenital malformations (MCM) | From date of conception (DOC) to pregnancy outcome for fetal losses or 12 months of infant age for live births
  Describe and estimate the risk of MCM in live and non-live offspring from the women who had moderate/severe SLE and were exposed to anifrolumab during the first trimester of pregnancy or exposed to SOC and unexposed to anifrolumab during the first trimester of pregnancy
Relative risk of MCM | From date of conception (DOC) to pregnancy outcome for fetal losses or 12 months of infant age for live births
  Estimate the relative risk of MCM in live and non-live offspring from the women who had moderate/severe SLE and were exposed to anifrolumab during the first trimester of pregnancy or exposed to SOC and unexposed to anifrolumab during the first trimester of pregnancy
Risk of select pregnancy loss outcomes | At delivery/birth
  Describe and estimate the risk of select pregnancy loss outcomes (composite of spontaneous abortion and stillbirth) in all pregnancies from women who had moderate/severe SLE and were exposed or unexposed to anifrolumab during pregnancy
Relative risk of select pregnancy loss outcomes | At delivery/birth
  Estimate the relative risk of select pregnancy loss outcomes (composite of spontaneous abortion and stillbirth) in pregnancies from women who had moderate/severe SLE and were exposed or unexposed to anifrolumab during pregnancy

SECONDARY OUTCOMES:
Demographic and clinical characteristics | From date of conception (DOC) to pregnancy outcome for fetal losses or 12 months of infant age for live births
  Describe the demographic and clinical characteristics of the live and non-live offspring and their mothers who had moderate/severe SLE and were exposed or unexposed to anifrolumab during the first trimester of pregnancy or anytime during pregnancy
Risk of minor congenital malformations (mCM) | From date of conception (DOC) to pregnancy outcome for fetal losses or 12 months of infant age for live births
  Describe and estimate the risk of mCM in live and non-live offspring from women with moderate/severe SLE who were exposed or unexposed to anifrolumab during pregnancy
Relative risk of mCM | From date of conception (DOC) to pregnancy outcome for fetal losses or 12 months of infant age for live births
  Estimate the relative risk of mCM in live and non-live offspring from women who had moderate/severe SLE and were exposed or unexposed to anifrolumab during pregnancy
Risk of adverse pregnancy outcomes | At delivery/birth
  Describe and estimate the risk of adverse pregnancy outcomes (ectopic pregnancy, spontaneous abortion, elective termination of pregnancy, stillbirth, infections requiring hospitalisation during pregnancy, emergency caesarean section) in all pregnancies from women who had moderate/severe SLE and were exposed or unexposed to anifrolumab during pregnancy
Relative risk of adverse pregnancy outcomes | At delivery/birth
  Estimate the relative risk of adverse pregnancy outcomes (ectopic pregnancy, spontaneous abortion, elective termination of pregnancy, stillbirth, infections requiring hospitalisation during pregnancy, emergency caesarean section) in pregnancies from women who had moderate/severe SLE and were exposed or unexposed to anifrolumab during pregnancy
Risk of adverse birth outcomes | At delivery/birth
  Describe and estimate the risk of adverse birth outcomes (preterm birth,
  small for gestational age (SGA)) in live offspring from women who had moderate/severe SLE and were exposed or unexposed to anifrolumab during pregnancy
Relative risk of adverse birth outcomes | At delivery/birth
  Estimate the relative risk of adverse birth outcomes (preterm birth, small for gestational age (SGA)) in live offspring from women who had moderate/severe SLE and were exposed or unexposed to anifrolumab during pregnancy

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/